CLINICAL TRIAL: NCT01378598
Title: Enhancing Adherence and Knowledge of Erlotinib in Patients Wtih Non-Small Cell Lung Cancer: A Feasibility Pilot Study
Brief Title: Enhancing Adherence and Knowledge of Erlotinib in Patients Wtih Non-Small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Joan Lucca, RN, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-171
Record Dates: First submitted 2010-12-27; First posted 2011-06-22 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Lung Cancer
Keywords: erlotinib; educational intervention; direct care nurse
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Nursing Educational Intervention — Four educational sessions with the direct care nurse (DCN)

SUMMARY:
Research has found that patients sometimes have trouble obtaining oral (by mouth) cancer medications, understanding how to take these pills, handling side effects related to these drugs, and remembering to take these medications. The purpose of this research study is to have direct care nurses (DCNs) in the Thoracic Oncology Program (TOP) clinic provide teaching and follow-up to patients starting erlotinib (using a teaching tool) and to test the feasibility of providing education and follow-up. This study will also evaluate if increasing knowledge about erlotinib helps participants manage side effects and stay on their erlotinib without interruptions.

DETAILED DESCRIPTION:
* Participants with non-small cell lung cancer will be asked to join this study after they have decided with their health care provider to start treatment with erlotinib (a pill).
* Educational Session 1 (Day that erlotinib is prescribed): During this clinic visit the physician or nurse practitioner will provide the participant with the DFCI Erlotinib Fact Sheet that reviews how to take the oral cancer medication and possible side effects to watch for. The TOP nurse will discuss the study and consent the participant. The TOP nurse will also provide participants with an Erlotinib Drug Log and instruct them on how use it to keep track of taking the erlotinib.
* Educational Session 2 (Within 72 hours of starting erlotinib): During this educational session, participants will talk with the TOP nurse by phone or in the clinic. The TOP nurse will use an oral cancer medication teaching tool (MOATT - Parts 1-4) to provide additional education about erlotinib. The MOATT tool was developed by the Multinational Association for Supportive Care in Cancer. This session will take about 20-30 minutes. Feasibility information will also be recorded by the nurse.
* Educational Session 3 (Phone follow-up 72 hours after Session 2): During this phone session, the TOP nurse will administer Parts 3-4 of the MOATT and discuss any side effects the participant is experiencing. This session will take 15-30 minutes. Feasibility information will also be documented.
* Educational Session 4 (First clinic visit after starting on Erlotinib): The TOP nurse will meet with the participant during their first DFCI clinic visit (with their physician or nurse practitioner), after starting erlotinib. During this session the participant will complete the Morisky Medication Adherence Scale 8-Item (MMAS-8), a Knowledge Rating Scale, and a demographic form. Parts 3-4 of the MOATT will also be administered, the Erlotinib Drug Log will be collected, and side effects will be discussed/recorded. This meeting will add 30-40 minutes to the clinic visit.
* After the participant completes Educational Session 4, their participation in the study will end.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Non-small cell lung cancer diagnosis
* Patient/provider decision to start erlotinib monotherapy
* No prior treatment with erlotinib
* Willingness to follow the protocol visit schedule
* Ability to understand and converse in English
* No major physical or psychological limitation that would interfere with study participation
* Not participating in other studies involving nurse/patient interactions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of a DCN educational intervention to enhance participant knowledge | 1 year
  To test the feasibility of direct care nurse (DCN) educational intervention to enhance participant knowledge of erlotinib and improve patient-reported adherence with regard to: 1) enrollment and retention rates, 2) DCN availability, 3) Completion of educational sessions and 4) Resources used or required for each session

SECONDARY OUTCOMES:
Describe the knowledge of and adherence to erlotinib as an oral anticancer agent | 1 year
  To describe the knowledge of (by MOATT) and adherence to (by MMAS 8-item) erlotinib as an oral anticancer agent in thoracic oncology patients.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Lucca, RN, MSN, NP-C, AOCN, Principal Investigator — Dana-Farber Cancer Institute